CLINICAL TRIAL: NCT06085794
Title: Comparative Study Between Standard PCNL and Endoscopic Combined Intrarenal Surgery (ECIRS) in the Galdakaomodified Supine Valdivia (GMSV) Position for Complex Nephrolithiasis in Obese Patients
Brief Title: Standard PCNL Vs Endoscopic Combined Intrarenal Surgery (ECIRS) for Complex Nephrolithiasis in Obese Patients
Acronym: ECIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Moataz bellah Mohamed, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECIRS complex stones in obese
Record Dates: First submitted 2023-09-13; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Renal Stone
Keywords: ECIRS; PCNL; Obese
MeSH Terms: conditions — Nephrolithiasis; Obesity | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Who Masked: Participant
Masking Description: 1st patient in the PCNL group , 2nd patient in ECIRS group and so on .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous nephrolithotomy (Active Comparator): the standard-PCNL group (will be performed by urologists with more than 2 years of experience of PCNL), Fluoroscopic-guided percutaneous renal access will be done for patients in the prone position.
  Interventions: Procedure: Percutaneous nephrolithotomy
- Endoscopic combined intrarenal surgery (Active Comparator): the ECIRS group (will be performed by urologists with more than 2 years of experience of PCNL and RIRS), patients will be oriented in the GMSV position.flexible ureteroscope will be inserted through the access sheath to observe the stone distributions. Under the guidance of fluoroscopy and endoscopic vision, a 18-20 Fr percutaneous tract will be established using sequential fascial dilators and a matching sheath for stone manipulation simultaneously. We use a 12-F nephroscope (Karl Storz).
  Interventions: Procedure: Endoscopic combined intrarenal surgery

INTERVENTIONS:
Procedure: Endoscopic combined intrarenal surgery — Combined complex stone clearance with mini-nephroscope and flexible URS
  Other Names: ECIRS
  Arms: Endoscopic combined intrarenal surgery
Procedure: Percutaneous nephrolithotomy — Clearance of renal stone with nephroscope in prone position
  Other Names: PCNL
  Arms: Percutaneous nephrolithotomy

SUMMARY:
Primary aim: comparing the efficacy of standard PCNL and endoscopic combined intrarenal surgery (ECIRS) in the Galdakao-modified Supine Valdivia (GMSV) position in a single session for the treatment of complex nephrolithiasis in obese patients.

Secondary aim: comparing safety and complications of standard PCNL and ECIRS in the GMSV.

DETAILED DESCRIPTION:
Complex nephrolithiasis including multiple peripheral or branched (partial or complete staghorn calculi) renal stones, is still currently an intractable problem for urologists to achieve stone-free status and minimize complication rates. According to the European Association of Urology Urolithiasis Guidelines, retrograde intrarenal surgery (RIRS) is recommended as first-line treatment for renal stones < 2 cm, and percutaneous nephrolithotomy (PCNL) is recommended as the gold standard for renal stones ≥ 2 cm in length.

Obesity has been identified as an independent risk factor for stone formation in the United States. Obesity (BMI >35) also places surgical patients at a greater risk of complications, because of the increased incidence in this group of diabetes, hypertension, ischemic heart disease, postoperative deep venous thrombosis, and pulmonary embolism, and because of poor radiographic visualization, obscure anatomic landmarks, more difficult renal access, and inferior stone-free rates.

Standard percutaneous nephrolithotomy (PCNL) is the recommended treatment by major guidelines. However, multiple tracts or sessions of PCNL were required to obtain a high stone-free rate (SFR) for complex renal calculi, especially staghorn stones, while procedure-related complications increased concomitantly. To acquire a higher SFR, full access to the entire intrarenal collecting system is the final goal of treatment for these patients suffering from multiple calyceal or peripheral satellite calculi, which is technically challenging by means of RIRS or PCNL monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Partial or complete staghorn stones)
* Guy's Stone Score III or IV)
* Adult (18-60) years old patients
* Obese & super-obese patients (BMI > 30 kg/m 2).

Exclusion Criteria:

* Patients with congenital renal anomalies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PCNL vs ECIRS | 2 days
  Operative duration in minutes (from positioning to the end of the procedure) will be recorded for the two groups Stone-free status will be evaluated with a plain abdominal radiograph of the kidneys, ureters, and bladder (KUB) for radiopaque stones and NCCT for lucent stones before hospital discharge. Stone-free status is defined as no or small calyceal residuals of ≤ 4 mm (clinically insignificant residual fragment) without infection.

SECONDARY OUTCOMES:
Safety and complication of PCNL Vs ECIRS | 1 month.
  Intraoperative complications will be recorded and 30-day postoperative complications will be graded according to the modified Clavien classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Liu YH, Jhou HJ, Chou MH, Wu ST, Cha TL, Yu DS, Sun GH, Chen PH, Meng E. Endoscopic Combined Intrarenal Surgery Versus Percutaneous Nephrolithotomy for Complex Renal Stones: A Systematic Review and Meta-Analysis. J Pers Med. 2022 Mar 28;12(4):532. doi: 10.3390/jpm12040532. PMID 35455648
- [Background] Cracco CM, Scoffone CM. ECIRS (Endoscopic Combined Intrarenal Surgery) in the Galdakao-modified supine Valdivia position: a new life for percutaneous surgery? World J Urol. 2011 Dec;29(6):821-7. doi: 10.1007/s00345-011-0790-0. Epub 2011 Nov 6. PMID 22057344
- [Background] Cracco CM, Scoffone CM. Endoscopic combined intrarenal surgery (ECIRS) - Tips and tricks to improve outcomes: A systematic review. Turk J Urol. 2020 Nov;46(Supp. 1):S46-S57. doi: 10.5152/tud.2020.20282. Epub 2020 Aug 25. PMID 32877638
- [Background] Grosso AA, Sessa F, Campi R, Viola L, Polverino P, Crisci A, Salvi M, Liatsikos E, Feu OA, DI Maida F, Tellini R, Traxer O, Cocci A, Mari A, Fiori C, Porpiglia F, Carini M, Tuccio A, Minervini A. Intraoperative and postoperative surgical complications after ureteroscopy, retrograde intrarenal surgery, and percutaneous nephrolithotomy: a systematic review. Minerva Urol Nephrol. 2021 Jun;73(3):309-332. doi: 10.23736/S2724-6051.21.04294-4. Epub 2021 Apr 22. PMID 33887891
- [Background] Knoll T, Daels F, Desai J, Hoznek A, Knudsen B, Montanari E, Scoffone C, Skolarikos A, Tozawa K. Percutaneous nephrolithotomy: technique. World J Urol. 2017 Sep;35(9):1361-1368. doi: 10.1007/s00345-017-2001-0. Epub 2017 Jan 25. PMID 28124111
- [Derived] Tawfeek AM, Higazy A, Elkenany MM, Taema K, Arafa H. Mini-Endoscopic Combined Intrarenal Surgery vs Percutaneous Nephrolithotomy in the Management of Complex Nephrolithiasis: A Randomized Controlled Trial. J Endourol. 2025 Oct;39(10):998-1004. doi: 10.1177/08927790251360265. Epub 2025 Jul 18. PMID 40681329